CLINICAL TRIAL: NCT01960543
Title: Comparison of the Effects of Bupivacaine or Levobupivacaine on Cerebral Oxygenation During Intrathecal Anesthesia in Elderly Patients Who Underwent Hip Fracture Repair
Brief Title: Effects of Bupivacaine and Levobupivacaine on Cerebral Oxygenation During Intrathecal Anesthesia in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Diana L Fernandez Galinski, Physician - Anesthesiology, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANE-INTRA-2013
Record Dates: First submitted 2013-09-23; First posted 2013-10-10 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Complication of Anesthesia
Keywords: Intrathecal anesthesia; Levobupivacaine; Bupivacaine; Hip fracture
MeSH Terms: conditions — Hip Fractures | interventions — Bupivacaine; Levobupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): Intrathecal administration of bupivacaine 0.5%
  Doses:
  Bupivacaine 7 mg plus fentanyl 15 ug for patients shorter than 160 cm. Bupivacaine 9 mg plus fentanyl 15 ug for patients equal or taller than 160 cm or hip replacement.
  Interventions: Drug: fentanyl 15 microg; Drug: Bupivacaine 7 mg; Drug: Bupivacaine 9 mg
- Levobupivacaine (Active Comparator): Intrathecal administration of levobupivacaine 0.5%:
  Doses:
  Levobupivacaine 7 mg plus fentanyl 15 ug for patients shorter than 160 cm. Levobupivacaine 9 mg plus fentanyl 15 ug for patients equal or taller than 160 cm or hip replacement.
  Interventions: Drug: fentanyl 15 microg; Drug: Levobupivacaine 7 mg; Drug: Levobupivacaine 9 mg

INTERVENTIONS:
Drug: fentanyl 15 microg
Drug: Bupivacaine 7 mg
  Arms: Bupivacaine
Drug: Bupivacaine 9 mg
  Arms: Bupivacaine
Drug: Levobupivacaine 7 mg
  Arms: Levobupivacaine
Drug: Levobupivacaine 9 mg
  Arms: Levobupivacaine

SUMMARY:
Elderly patients with hip fracture are frail due to associated comorbidity. In these situations, regional anesthesia is recommended as it is associated to less postoperative cognitive dysfunction. However, hypotension during the process may impair ischemic cardiopathy and induce a cerebrovascular stroke. Selection of the right anesthetic agent and the administration of vasoactive drugs during the process can minimize these risks. Although bupivacaine and levobupivacaine share pharmacokinetic and pharmacodynamic properties, the studies show conflicting results. The aim of this study is to investigate if there are clinically relevant differences between these two drugs in terms of hemodynamic parameters during the surgical process with special focus on the effects on regional cerebral oximetry and cognitive status after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 70 years old who undergo major surgery for hip fracture and will receive intrathecal anesthesia
2. Patients in which it is considered adequate, according to the usual clinical practice, the use of bupivacaine or levobupivacaine as part of the intrathecal anesthesia
3. Patients who give their informed consent to participate in the study

Exclusion Criteria:

1. Patients allergic to anesthetic drugs to be used in the protocol or to local anesthetics amida type.
2. Patients with severe aortic stenosis or hemodynamic instability.
3. Patients who refuse the anesthetic technique or contraindication for the use of the intrathecal technique.
4. Patients with severe cognitive impairment previous to the intervention (defined by a score in the Pfeiffer test of 8-10 errors)
5. Patients in which the use of bupivacaine or levobupivacaine is contraindicated as part of the intrathecal anesthesia
6. Any condition that, in the investigator's opinion, could pose a risk to the patient

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of intraoperative time with a decrease of cerebral regional oxygen saturation (SrO2), of at least 20% with respect to baseline values | Measured continuously during surgery (an expected average of 60 minutes)

SECONDARY OUTCOMES:
Change in cognitive function after 7 days with respect to preoperative function, measured by means of the Pfeiffer cognitive test | 7 days post surgery

OTHER OUTCOMES:
Proportion of intraoperative time with a decrease in values of cerebral regional oxygen saturation to 40% or 50% | Measured continuously during surgery (an expected average of 60 minutes)
Time to first drop of cerebral regional oxygen saturation below 40% or 50% | Assessed up to the end of surgery (an expected average of 60 minutes)
Changes in cerebral regional oxygen saturation induced by the administration of vasoconstrictor drugs | Measured continuously for the whole duration of surgery (an expected average of 60 minutes)
Doses of vasoactive drugs administered | measured up to the end of surgery (an expected average of 60 minutes)
Adverse events and mortality | 30 days
Blood pressure | Measured continuously for the whole duration of surgery (an expected average of 60 minutes)
Heart Rate | Measured continuously for the whole duration of surgery (an expeted average of 60 minutes)
Oxygen saturation during the surgery | Measured continuously for the whole duration of surgery (an expected average of 60 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Sabadell, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Vives R, Fernandez-Galinski D, Gordo F, Izquierdo A, Oliva JC, Colilles C, Pontes C. Effects of bupivacaine or levobupivacaine on cerebral oxygenation during spinal anesthesia in elderly patients undergoing orthopedic surgery for hip fracture: a randomized controlled trial. BMC Anesthesiol. 2019 Jan 31;19(1):17. doi: 10.1186/s12871-019-0682-1. PMID 30704463